CLINICAL TRIAL: NCT01263002
Title: An Open Study to Evaluate the Efficacy, Safety and Sustained Effect of Clevudine Monotherapy or Adefovir and Clevudine Combination in Proportion to Roadmap Concept in Patients With Chronic Hepatitis B Associated Hepatocellular Carcinoma
Brief Title: A Study With Clevudine Monotherapy or Adefovir and Clevudine Combination in Proportion to Roadmap Concept in Patients With HBV Associated-HCC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bukwang Pharmaceutical (Industry)
Responsible Party: Myunghyun Jeong, Bukwang
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLV-413
Record Dates: First submitted 2010-12-17; First posted 2010-12-20 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Hepatitis B Associated Hepatocellular Carcinoma
MeSH Terms: interventions — clevudine; adefovir

INTERVENTIONS:
Drug: clevudine, Adefovir — Nucleoside-analogue naive patient : Clevudine 30mg qd
  1. Assess the complete virological response(HBV DNA < 60 IU/ml) at 24 weeks: Only Clevudine 30mg qd
  2. Assess not the complete virological response at 24 weeks : Add Adefovir 10mg qd
  3. During medication of Clevudine, virological breakthrough : add adefovir 10mg qd
  4. During treatment period, composite virological response : stop the medication and F/U for 2 years
  5. Recurrence after stopping treatment(HBV DNA > 2,000IU/ml) retreat medication at composite virological response.
     * complete virological response: HBV DNA < 60 IU/ml
     * virological breakthrough : During antiviral treatment, HBV DNA increased from nadir to 1 log10IU/ml continuously.

SUMMARY:
An open study to evaluate the Efficacy, Safety of Clevudine monotherapy or Adefovir and Clevudine combination in Proportion to Roadmap Concept in patients with chronic hepatitis B Associated Hepatocellular Carcinoma

ELIGIBILITY:
Inclusion Criteria

1. Patient with chronic HBV DNA and/or with symptoms of liver cirrhosis
2. Patient with Hepatocellular carcinoma evidenced by sonography, CT scan, or MRI scan)
3. Patient is 18 years and older.
4. Patient is documented to be HBsAg positive for > 6 months.

   * Laboratory report proving HBsAg positive or HBeAg positive for at least six months
   * IgM anti-HBc negative, IgG anti-HBc positive at screening
5. Patient is HBV DNA positive with DNA levels ≥ 2,000 IU/mL within 30 days of baseline.
6. Patient has ALT or AST levels >=40 IU/L
7. Cell carcinoma/hepatocellular carcinoma patient who is anticipated to live at least 1 year.
8. Patient who is fully active, able to carry on all pre-disease performance without restriction or restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
9. Patient who is classified as NYHA functional classification grade 1-2. (NYHA;New York Heart Association)
10. Patient who is able to give written informed consent prior to study start and to comply with the study requirements.

Exclusion Criteria

1. Patient is currently receiving antiviral therapy.
2. Patients previously treated with interferon, peg-interferon or other immunomodulatory within the previous 6 months.
3. Patients previously treated with clevudine, lamivudine, adefovir, entecavir, telbivudine, tenofovir or any other investigational nucleoside for HBV infection.
4. Patient is coinfected with HCV, HDV or HIV.
5. Patient with metastatic malignancy.
6. Patient with previous liver transplantation
7. Patient is pregnant or breast-feeding.
8. Patient has a clinically relevant history of abuse of alcohol or drugs.
9. Patient use oriental medicine within the previous 2 weeks.
10. Patient has a significant immunocompromised, gastrointestinal, renal, hematological, psychiatric, bronchopulmonary, biliary diseases excluding asymptomatic GB stone, neurological, cardiac, oncologic(except HCC)or allergic disease or medical illness that in the investigator's opinion might interfere with therapy.
11. Patient has creatinine clearance less than 60mL/min as estimated by the following formula: (140-age in years) (body weight [kg])/(72) (serum creatinine [mg/dL]) [Note: multiply estimates by 0.85 for women]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2010-06; Primary Completion 2013-01 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with HBV DNA levels < 60 IU/mL | 48 week

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea